CLINICAL TRIAL: NCT05186428
Title: Evaluation of a Non-invasive Urinary Collection Technique for the Adaptation of Diuretic Treatment in Incontinent Heart Failure Patient Over 75 Years of Age in the Acute Phase
Acronym: ATIICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATIICA
Record Dates: First submitted 2021-12-03; First posted 2022-01-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diuresis in Incontinent Patients
MeSH Terms: interventions — Diapers, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The "before" period (Other)
  Interventions: Other: carrying out standard care
- the "after" period (Experimental)
  Interventions: Other: adult diaper

INTERVENTIONS:
Other: carrying out standard care — The adaptation of the diuretic treatment will be made according to the possible diuresis records and the weighing of the patient every 2 days.
  Arms: The "before" period
Other: adult diaper — the diuresis which will be calculated by making the difference between the weight of the soiled protection weighed and the weight of the dry protection
  Arms: the "after" period

SUMMARY:
Heart failure is a general disease affecting many organs and regulatory systems with a prevalence of 10% after 75 years of age, leading to significant hospitalization in the elderly. This generates a significant cost for our health system. The management of patients over 75 years of age in acute heart failure requires special monitoring of diuresis and weight. However, it is sometimes difficult to collect urine from incontinent elderly patients (not catheterized, habitually wearing protection) under intravenous diuretics. The evaluation of a non-invasive technique of urine collection for the adaptation of diuretic treatment in the incontinent patient with heart failure over 75 years of age in the acute phase seems to us to be interesting to conduct.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 75 years of age
* Geriatric short-stay inpatient, geriatric/cardio medicine unit geriatrics
* Incontinent patient with urinary protection
* Patient with acute heart failure according to the diagnosis made by the doctors of unity
* Patient treated with intravenous diuretic
* Patient benefiting from a social security scheme or benefiting from it by a third party
* Patient who gave their non-opposition to the study after clear information

Exclusion Criteria:

* Patient hospitalized in another unit of the geriatric division
* Patient allergic to the protections provided
* Patient carrying a bladder probe upon entry into the unit
* Patient with a precarious non-perfusable venous capital

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of the duration of intravenous diuretic treatment during 2 periods | 15 days maximum
  The duration of intravenous diuretic treatment in incontinent heart failure patients over 75 years old without urinary catheterization during 2 period (before and after)
  * Before" period with usual diuresis measurement
  * After" period with weighing of diapers

SECONDARY OUTCOMES:
Comparison comfort of patient between the 2 periods with VAS | 15 days maximum
Compare between the 2 periods the rate of skin complications related to the 2 diuresis assessment techniques, | 15 days maximum
Compare between the 2 periods the rate of bladder catheterization during the study | 15 days maximum
Compare the mortality rate between the 2 periods | 15 days maximum
Compare the average length of stay of patients between the 2 periods | 15 days maximum

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PAJOUX, Principal Investigator — CHU de Poitiers FRANCE
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided